CLINICAL TRIAL: NCT04302116
Title: Efficacy of Vigabatrin With High Dose Prednisolone Combination Therapy Versus Vigabatrin Alone for Infantile Spasm: a Randomized Trial
Brief Title: Vigabatrin With High Dose Prednisolone Combination Therapy vs Vigabatrin Alone for Infantile Spasm
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kullasate Sakpichaisakul (Other Government)
Responsible Party: Sponsor-Investigator, Kullasate Sakpichaisakul, Pediatric epileptologist, Queen Sirikit National Institute of Child Health
Organization: Queen Sirikit National Institute of Child Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QSNICH63-008
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Infantile Spasm; West Syndrome
Keywords: Infantile Spasm; Vigabatrin; Prednisolone; Treatment; West Syndrome
MeSH Terms: conditions — Spasms, Infantile | interventions — Combined Modality Therapy; Vigabatrin; Prednisolone

STUDY DESIGN:
Intervention Model Description: A pragmatic parallel group randomised trial comparing vigabatrin with high dose prednisolone to vigabatrin treatment alone in the treatment of infantile spasm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Each patient will visit the clinic at Day 8, 14, 43, and 3 months by outcome assessor who is blinded for treatment to determine seizure frequency and adverse events. Those patients will be seen and under taking care of primary neurologists and pharmacists who are not blinded to treatment at the same visit as a standard clinical practice and check with compliance and adjust vigabatrin or prednisolone following each treatment allocated (if needed). Family or caregivers will not be blinded to treatment. EEG will be scored using BASED scores at Day 0 (before treatment), 14, and 43 to assess the resolution of hypsarrhythmia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination therapy with vigabatrin and prednisolone (Experimental): Vigabatrin (tablet of 500 mg) dose based on weight divided in two times. The protocol for vigabatrin dose is 50 mg/kg/day at Day 1, 100 mg/kg/day at Day 2, and increase to 150 mg/kg/day if seizures still occur after 72 hours after treatment. Vigabatrin will be continued for 3 months, then reduced and completely off within 4 weeks.
  Prednisolone (tablet of 5 mg), 40 mg of prednisolone (10 mg oral 4 times a day) for 14 days. Prednisolone will be increased to 60 mg/day (20 mg oral 3 times a day) if seizures still occur at Day 7 or recur within Day 8 - 14. Then, prednisolone will be reduced every 5 day until completely off within 1 month. Total prednisolone duration is 1 month.
  Interventions: Drug: Combination therapy with vigabatrin and prednisolone
- Vigabatrin alone (Active Comparator): Vigabatrin (500 mg/tab) dose will be calculated on weight basis divided in two times. The protocol for vigabatrin dose is 50 mg/kg/day at Day 1, 100 mg/kg/day at Day 2, and increase to 150 mg/kg/day if seizures still occur after 72 hours after treatment.
  Vigabatrin will be continued for 3 months, then reduced and completely off within 4 weeks.
  Interventions: Drug: Vigabatrin Tablets

INTERVENTIONS:
Drug: Combination therapy with vigabatrin and prednisolone — High dose prednisolone (40 - 60 mg/day) for 1 month combined with vigabatrin treatment (50-150 mg/kg/day) twice daily for 4 months
  Other Names: Sabril with prednisolone
  Arms: Combination therapy with vigabatrin and prednisolone
Drug: Vigabatrin Tablets — Vigabatrin (50-150 mg/kg/day) twice daily for 4 months
  Other Names: Sabril
  Arms: Vigabatrin alone

SUMMARY:
Infantile spasms (IS) are seizures associated with a severe infantile epileptic encephalopathy. Both cessation of spasms and electrographic response are necessary for the best neurodevelopmental outcomes. Adrenocorticotrophic hormone (ACTH), or prednisolone, or vigabatrin are considered the first-line treatment individually. However, ACTH expense and availability are the barriers in developing countries including Thailand. Vigabatrin, therefore, is the first recommended by Epilepsy Society of Thailand due to ACTH unavailability. Recently, combined steroid treatments (either ACTH or high dose prednisolone) with vigabatrin are superior in cessation of spasms compared to steroid treatment alone. Thus, this study is aimed to compare the efficacy of vigabatrin with high dose prednisolone combination therapy and vigabatrin alone.

DETAILED DESCRIPTION:
Infantile spasms are recognized as epileptic encephalopathy which include the hypsarrhythmia or variants electroencephalographic (EEG) features and psychomotor regression. Various underlying conditions are associated with the infantile spasm included cerebral malformation, hypoxic ischemic encephalopathy, genetic disorders (Down syndrome), tuberous sclerosis complex (TSC), etc. Although vigabatrin has the evidence to use as the first line treatment for infantile spasm related with TSC. Adrenocorticotrophic hormone (ACTH), or high dose prednisolone, or vigabatrin are the first line treatment of IS in non-TSC.

The effectiveness of ACTH versus high dose prednisolone question have not yet definitely answered. Furthermore, ACTH expense and availability are the barriers in developing countries including Thailand. Vigabatrin, therefore, is the first option of therapy recommended by Epilepsy Society of Thailand due to ACTH unavailability. Recently, combined steroid treatments (either ACTH or high dose prednisolone) with vigabatrin are superior in cessation of spasms compared to steroid treatment alone. Questions about the clinical cessation of IS and electrographic remission by combination treatment with vigabatrin and high dose prednisolone compare to vigabatrin alone have not fully elucidated. Thus, this study is aimed to compare the efficacy of vigabatrin with high dose prednisolone combination therapy and vigabatrin alone.

ELIGIBILITY:
Inclusion Criteria:

* Age at 2-14 months at date of enrollment
* Clinical diagnosis of infantile spasm assessed by pediatric neurologist and hypsarrhythmic pattern or variants interpreted by pediatric epileptologist
* Thai nationality

Exclusion Criteria:

* Previous treatment (within the last 28 days) with vigabatrin or corticosteroid
* Previous diagnosis of epileptic encephalopathy e.g. early infantile epileptic encephalopathy and early myoclonic epileptic encephalopathy
* Has a clinical suspicious or diagnosis of tuberous sclerosis complex characterized by one of these; known affected parent, previously diagnosed cardiac rhabdomyoma, hypomelanotic macules, forehead fibrous plaque, shagreen patch, retinal phakoma, or known polycystic kidneys
* A contraindication to vigabatrin or corticosteroid such as recent varicella or herpes zoster infection, gastrointestinal hemorrhage etc.
* Thai language ability of the parents or guardians is that they may not understand what is being requested of them.
* Predictable lack of availability of follow up

Ages: 2 Months to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Cessation of spasms | Assessed during Day 14 to Day 42 after treatment.
  Defined as no witnessed spasms (either clusters or single spasms) from Day 14 to Day 42 inclusive.

SECONDARY OUTCOMES:
Electrographic response | Assessed during Day 14 and Day 43 after treatment.
  Disappearance of hypsarrhythmia defined by Burden of Amplitudes and Epileptiform Discharges (BASED) scoring system < 2 at Day 14 and Day 43 after treatment.
Electroclinical response | Between Day 14 and Day 21.
  the cessation of spasms with the addition of absence of hypsarrhythmia (BASED score < 2) on the Day 14 EEG. Valid Day 14 EEGs will be undertaken between Day 14 and Day 21 inclusive.
Extended electroclinical response | Between Day 42 and Day 49.
  Electroclinical response with the addition of absence of hypsarrhythmia (BASED score < 2) on the Day 42 EEG. Valid Day 42 EEGs will be undertaken between Day 42 and Day 49 inclusive.
The time taken to absence of spasms | Day 1 to Day 14
  Duration for clinical cessation of spasms after initiation treatment
Relapse of spasms | Day 42 to 3 months after treatment
  Defined when a cluster of more than one spasm in reported after Day 42. No EEG is required.
Adverse reactions | Day 1 to Day 14, from Day 15 to Day 42, and from Day 43 to 4 months into the trial
  Each adverse event will be evaluated by the principal investigator to determine whether in their view it is an adverse reaction. If considered an adverse reaction, it will be reported by using the standard classification.
Epilepsy outcome at age 18 months | From Day 42 to age 18 months
  Epilepsy status and antiepileptic drugs (AEDs) will be recorded by using the following categories: 1) Infantile spasms (clusters of spasms), 2) Any other epileptic seizure including febrile seizures, and 3) Names of any preventive AEDs prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Kullasate Sakpichaisakul, MD, Principal Investigator — Queen Sirikit National Institute of Child Health
Locations (1):
- Queen Sirikit National Institute of Child Health, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available for the confidentiality.

REFERENCES:
- [Result] Hrachovy RA, Frost JD Jr. Infantile epileptic encephalopathy with hypsarrhythmia (infantile spasms/West syndrome). J Clin Neurophysiol. 2003 Nov-Dec;20(6):408-25. doi: 10.1097/00004691-200311000-00004. PMID 14734931
- [Result] Jeavons PM, Bower BD, Dimitrakoudi M. Long-term prognosis of 150 cases of "West syndrome". Epilepsia. 1973 Jun;14(2):153-64. doi: 10.1111/j.1528-1157.1973.tb03952.x. No abstract available. PMID 4515986
- [Result] Trevathan E, Murphy CC, Yeargin-Allsopp M. The descriptive epidemiology of infantile spasms among Atlanta children. Epilepsia. 1999 Jun;40(6):748-51. doi: 10.1111/j.1528-1157.1999.tb00773.x. PMID 10368073
- [Result] Hrachovy RA, Frost JD Jr, Kellaway P. Hypsarrhythmia: variations on the theme. Epilepsia. 1984 Jun;25(3):317-25. doi: 10.1111/j.1528-1157.1984.tb04195.x. PMID 6539199
- [Result] Pellock JM, Hrachovy R, Shinnar S, Baram TZ, Bettis D, Dlugos DJ, Gaillard WD, Gibson PA, Holmes GL, Nordl DR, O'Dell C, Shields WD, Trevathan E, Wheless JW. Infantile spasms: a U.S. consensus report. Epilepsia. 2010 Oct;51(10):2175-89. doi: 10.1111/j.1528-1167.2010.02657.x. PMID 20608959
- [Result] Lux AL, Osborne JP. A proposal for case definitions and outcome measures in studies of infantile spasms and West syndrome: consensus statement of the West Delphi group. Epilepsia. 2004 Nov;45(11):1416-28. doi: 10.1111/j.0013-9580.2004.02404.x. PMID 15509243
- [Result] Mackay MT, Weiss SK, Adams-Webber T, Ashwal S, Stephens D, Ballaban-Gill K, Baram TZ, Duchowny M, Hirtz D, Pellock JM, Shields WD, Shinnar S, Wyllie E, Snead OC 3rd; American Academy of Neurology; Child Neurology Society. Practice parameter: medical treatment of infantile spasms: report of the American Academy of Neurology and the Child Neurology Society. Neurology. 2004 May 25;62(10):1668-81. doi: 10.1212/01.wnl.0000127773.72699.c8. PMID 15159460
- [Result] Wheless JW, Clarke DF, Arzimanoglou A, Carpenter D. Treatment of pediatric epilepsy: European expert opinion, 2007. Epileptic Disord. 2007 Dec;9(4):353-412. doi: 10.1684/epd.2007.0144. PMID 18077226
- [Result] Demarest ST, Shellhaas RA, Gaillard WD, Keator C, Nickels KC, Hussain SA, Loddenkemper T, Patel AD, Saneto RP, Wirrell E, Sanchez Fernandez I, Chu CJ, Grinspan Z, Wusthoff CJ, Joshi S, Mohamed IS, Stafstrom CE, Stack CV, Yozawitz E, Bluvstein JS, Singh RK, Knupp KG; Pediatric Epilepsy Research Consortium. The impact of hypsarrhythmia on infantile spasms treatment response: Observational cohort study from the National Infantile Spasms Consortium. Epilepsia. 2017 Dec;58(12):2098-2103. doi: 10.1111/epi.13937. Epub 2017 Nov 3. PMID 29105055
- [Result] Arya R, Shinnar S, Glauser TA. Corticosteroids for the treatment of infantile spasms: a systematic review. J Child Neurol. 2012 Oct;27(10):1284-8. doi: 10.1177/0883073812453203. Epub 2012 Aug 1. PMID 22859699
- [Result] Go CY, Mackay MT, Weiss SK, Stephens D, Adams-Webber T, Ashwal S, Snead OC 3rd; Child Neurology Society; American Academy of Neurology. Evidence-based guideline update: medical treatment of infantile spasms [RETIRED]. Report of the Guideline Development Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2012 Jun 12;78(24):1974-80. doi: 10.1212/WNL.0b013e318259e2cf. PMID 22689735
- [Result] Mytinger JR, Camfield PR. Synthetic ACTH Is Not Superior to Prednisolone for Infantile Spasms: Randomized Clinical Trials and Tribulations. Pediatr Neurol. 2015 Sep;53(3):181-2. doi: 10.1016/j.pediatrneurol.2015.07.005. Epub 2015 Jul 22. No abstract available. PMID 26302697
- [Result] Aicardi J, Mumford JP, Dumas C, Wood S. Vigabatrin as initial therapy for infantile spasms: a European retrospective survey. Sabril IS Investigator and Peer Review Groups. Epilepsia. 1996 Jul;37(7):638-42. doi: 10.1111/j.1528-1157.1996.tb00627.x. PMID 8681895
- [Result] Appleton RE, Peters AC, Mumford JP, Shaw DE. Randomised, placebo-controlled study of vigabatrin as first-line treatment of infantile spasms. Epilepsia. 1999 Nov;40(11):1627-33. doi: 10.1111/j.1528-1157.1999.tb02049.x. PMID 10565592
- [Result] Elterman RD, Shields WD, Mansfield KA, Nakagawa J; US Infantile Spasms Vigabatrin Study Group. Randomized trial of vigabatrin in patients with infantile spasms. Neurology. 2001 Oct 23;57(8):1416-21. doi: 10.1212/wnl.57.8.1416. PMID 11673582
- [Result] Maguire MJ, Hemming K, Wild JM, Hutton JL, Marson AG. Prevalence of visual field loss following exposure to vigabatrin therapy: a systematic review. Epilepsia. 2010 Dec;51(12):2423-31. doi: 10.1111/j.1528-1167.2010.02772.x. Epub 2010 Nov 10. PMID 21070215
- [Result] Lux AL, Edwards SW, Hancock E, Johnson AL, Kennedy CR, Newton RW, O'Callaghan FJ, Verity CM, Osborne JP. The United Kingdom Infantile Spasms Study comparing vigabatrin with prednisolone or tetracosactide at 14 days: a multicentre, randomised controlled trial. Lancet. 2004 Nov 13-19;364(9447):1773-8. doi: 10.1016/S0140-6736(04)17400-X. PMID 15541450
- [Result] Snead OC 3rd, Benton JW, Myers GJ. ACTH and prednisone in childhood seizure disorders. Neurology. 1983 Aug;33(8):966-70. doi: 10.1212/wnl.33.8.966. PMID 6308515
- [Result] Baram TZ, Mitchell WG, Tournay A, Snead OC, Hanson RA, Horton EJ. High-dose corticotropin (ACTH) versus prednisone for infantile spasms: a prospective, randomized, blinded study. Pediatrics. 1996 Mar;97(3):375-9. PMID 8604274
- [Result] Yi ZS, Wu HP, Yu XY, Chen Y, Zhong JM. Efficacy and tolerability of high-dose prednisone in Chinese children with infantile spasms. Brain Dev. 2015 Jan;37(1):23-8. doi: 10.1016/j.braindev.2014.02.005. Epub 2014 Mar 20. PMID 24657009
- [Result] Wanigasinghe J, Arambepola C, Sri Ranganathan S, Sumanasena S, Attanapola G. Randomized, Single-Blind, Parallel Clinical Trial on Efficacy of Oral Prednisolone Versus Intramuscular Corticotropin on Immediate and Continued Spasm Control in West Syndrome. Pediatr Neurol. 2015 Sep;53(3):193-9. doi: 10.1016/j.pediatrneurol.2015.05.004. Epub 2015 Jun 26. PMID 26216500
- [Result] O'Callaghan FJ, Edwards SW, Alber FD, Hancock E, Johnson AL, Kennedy CR, Likeman M, Lux AL, Mackay M, Mallick AA, Newton RW, Nolan M, Pressler R, Rating D, Schmitt B, Verity CM, Osborne JP; participating investigators. Safety and effectiveness of hormonal treatment versus hormonal treatment with vigabatrin for infantile spasms (ICISS): a randomised, multicentre, open-label trial. Lancet Neurol. 2017 Jan;16(1):33-42. doi: 10.1016/S1474-4422(16)30294-0. Epub 2016 Nov 10. PMID 27838190
- [Result] Ko A, Youn SE, Chung HJ, Kim SH, Lee JS, Kim HD, Kang HC. Vigabatrin and high-dose prednisolone therapy for patients with West syndrome. Epilepsy Res. 2018 Sep;145:127-133. doi: 10.1016/j.eplepsyres.2018.06.013. Epub 2018 Jun 23. PMID 29966811
- [Result] Mytinger JR, Hussain SA, Islam MP, Millichap JJ, Patel AD, Ryan NR, Twanow JD, Heyer GL. Improving the inter-rater agreement of hypsarrhythmia using a simplified EEG grading scale for children with infantile spasms. Epilepsy Res. 2015 Oct;116:93-8. doi: 10.1016/j.eplepsyres.2015.07.008. Epub 2015 Jul 28. PMID 26280806
- [Result] Kankirawatana P, Raksadawan N, Balangkura K. Vigabatrin therapy in infantile spasms. J Med Assoc Thai. 2002 Aug;85 Suppl 2:S778-83. PMID 12403260
- [Result] Visudtibhan A, Chiemchanya S, Visudhiphan P, Phusirimongkol S. Vigabatrin in infantile spasms: preliminary result. J Med Assoc Thai. 1999 Oct;82(10):1000-5. PMID 10561962
- [Derived] Boonkrongsak R, Trongkamolchai K, Suwannachote S, Sri-Udomkajorn S, Wittawassamrankul R, Arya R, Sakpichaisakul K. Combination Therapy With Vigabatrin and Prednisolone Versus Vigabatrin Alone for Infantile Spasms. Ann Clin Transl Neurol. 2025 May;12(5):1012-1021. doi: 10.1002/acn3.70034. Epub 2025 Mar 21. PMID 40116235
- See also: Clinical practice guidelines for epilepsy by Epilepsy Society of Thailand — http://thaiepilepsysociety.com/wp-content/uploads/2016/11/%E0%B9%81%E0%B8%99%E0%B8%A7%E0%B8%97%E0%B8%B2%E0%B8%87%E0%B9%80%E0%B8%A7%E0%B8%8A%E0%B8%9B%E0%B8%8F%E0%B8%B4%E0%B8%9A%E0%B8%B1%E0%B8%95%E0%B8%B4%E0%B9%82%E0%B8%A3%E0%B8%84%E0%B8%A5%E0%B8%A1%E0%B8%8A%E0%B8%B1%E0%B8%81%E0%B8%AA%E0%B8%B3%E0%B8%AB%E0%B8%A3%E0%B8%B1%E0%B8%9A%E0%B9%81%E0%B8%9E%E0%B8%97%E0%B8%A2%E0%B9%8C_2015.pdf